CLINICAL TRIAL: NCT01524874
Title: A Comparative Effectiveness Trial of High-quality Vitamin D3 Nutritional Supplements to Replete Serum Vitamin D
Brief Title: Comparative Effectiveness of Vitamin D and Repletion Strategies
Acronym: CEDARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bastyr University (Other)
Collaborators: Diabetes Action Research and Education Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H30-B11
Record Dates: First submitted 2011-11-08; First posted 2012-02-02 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Hypovitaminosis D; Insulin Resistance; Diabetes
Keywords: vitamin d; cholecalciferol; nutritional supplements; hypovitaminosis d; klotho; toll like receptor 4
MeSH Terms: conditions — Vitamin D Deficiency; Insulin Resistance; Diabetes Mellitus; Macular Degeneration, Age-Related, 10 | interventions — Cholecalciferol; Calcitriol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Powder D3 Capsule - 2,000 IU per Cap (Active Comparator): Vital Nutrients
  Interventions: Dietary Supplement: Vitamin D3
- Chewable D3 Tablet - 2,000 IU per Tab (Active Comparator): Integrative Therapeutics Inc.
  Interventions: Dietary Supplement: Vitamin D3
- Liquid D3 Drop - 2,000 IU per Drop (Active Comparator): Biotics Research
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 10,000 IU per Day for 12 Weeks
  Other Names: Calcitriol
  Arms: Powder D3 Capsule - 2,000 IU per Cap
Dietary Supplement: Vitamin D3 — 10,000 IU per Day for 12 Weeks
  Other Names: Calcitriol
  Arms: Chewable D3 Tablet - 2,000 IU per Tab
Dietary Supplement: Vitamin D3 — 10,000 IU per Day for 12 Weeks
  Other Names: Calcitriol
  Arms: Liquid D3 Drop - 2,000 IU per Drop

SUMMARY:
The importance of vitamin D (VitD) in the prevention and treatment of human health conditions has gained increased attention in recent years. As a result, medical providers of all categories are screening clinical VitD status frequently, yet become challenged with how to best advise patients regarding repletion of VitD status, i.e. which form of VitD replacement is most effective. It has been recognized that to achieve significant effects - serum concentrations >30ng/ml (75 nmol/ml) - it is necessary, as well as safe, to recommend substantially higher doses than were previously thought sufficient. These higher doses can be easily achieved orally. This clinical trial aims to compare absorption of three available forms of this fat-soluble vitamin, due to the potential differences in absorption of different preparations. High-quality powdered, chewable and lipid-emulsified VitD are readily available as supplements, yet these have not been systematically compared. This three-arm, randomized clinical trial will compare the difference in serum 25-hydroxycholecalciferol (25-OH)D concentration between the three arms at baseline and after random administration of one of the three VitD preparations for 12-weeks at a dosage of 10,000 IU VitD per day. The investigators hypothesize that the three forms of vitD will result in an equivalent increase in serum 25OHD.

DETAILED DESCRIPTION:
VitD has numerous hormonal effects, including regulation of Ca2+ and Mg2+, as well as effects on numerous genes, including insulin and androgens. Mounting literature demonstrates associations between VitD insufficiency and cancer, diabetes and heart disease. VitD insufficiency, defined by concentration of serum 25-hydroxycholecalciferol (25-OHD) <33ng/ml (82.5 nmol/ml), is common at all latitudes; the prevalence is estimated at ~35% in "healthy" populations. VitD testing and replacement is gaining popularity in clinical practice. It is not known whether there is a difference in the effect of equivalent doses of emulsified vs. non-emulsified cholecalciferol (VitD3) supplementation, reflected by quantitative changes in serum 25-OHD. However, clinical observations revealed that in an average of 4.4 months, subjects taking 4000 iu daily of the emulsified form of cholecalciferol improved their 25-OHD levels by 6.76 ng/mL more than those taking 5,000 iu daily of the non-emulsified form. The safety of taking 10,000 IU/day has been confirmed. Taking this dose for 12 weeks should cause a robust increase in serum 25-OHD. This study will provide preliminary data comparing three high quality VitD3 supplements, one a powdered capsule, one a chewable tablet, and the other a lipid-emulsified liquid. Future studies will compare the "better" supplement to conventional VitD replacement using VitD2.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Between18-65 years of age; there is an age-related decline in the absorption, transport or liver hydroxylation of orally-consumed VitD (Harris, 1999) therefore adults older than 65 will be excluded. This population is also at greater risk of being on medications with potential medication interactions, e.g. anticoagulants.
* Willingness to perform baseline screening tests: serum 25-OHD, CBC, Comprehensive metabolic chemistry panel (electrolytes, hepatic and renal function tests, lipids, HgA1C, insulin and glucose)
* Screening serum 25-OHD <33ng/ml (82.5 nmol/ml). If >=33ng/ml (82.5 nmol/ml), subjects will participate in the research study as baseline controls for the nested studies of Klotho and TLR-4.
* Ability to read and speak English
* Willingness to be randomized to one of three active treatments for 3 months

Exclusion Criteria:

* Subjects who have a serum baseline 25-OHD >=33ng/ml (82.5 nmol/ml) will be excluded once the VitD sufficient baseline control recruitment goal is met
* Subjects who have historical or current use of extra-dietary VitD, other than what is in a multivitamin, for the previous 3 months.
* LFTs: AST>60 U/L; ALT>65 U/L; Alkaline phosphatase >120 U/L. Total bilirubin>1.5 mg/dL
* Serum creatinine>1.4 mg/dL; BUN >25 mg/dL5. Subjects who are pregnant, or could become pregnant, unless they are using regular birth control (OCPs, condoms, IUD).
* Subjects who have established osteoporosis.
* Subjects who have history or symptoms of a parathyroid disorder.
* Subjects who have difficulty swallowing pills.
* Subjects who are unwilling to use sunscreen.
* Subjects who have had a past adverse reaction to sunscreen.
* Subjects who are taking medications over the previous 3 months that interfere with the metabolism of VitD (anti-convulsants, anti-coagulants, oral corticosteroids, or barbiturates).
* Subjects with any psychological conditions or substance abuse that may make the subject non- adherent, such as history of bipolar disorder, mania, untreated anxiety or other mood disorder, as determined by the site PI.
* Other severe illness or mental incapacity that, in the opinion of the site PI, would render the potential subject incapable of participating in the study.
* Allergy to sesame oil base
* Heart arrhythmia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-08; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change in mean serum 25-hydroxycholecalciferol concentration | Baseline and 12 weeks
  To compare the change in serum 25-hydroxycholecalciferol (25-OHD) concentration between three forms of supplemental vitamin D3: a lipid-emulsified form administered in a sesame oil base, a non-emulsified chewable tablet, and a non-emulsified form administered as a capsule, following 12 weeks of supplementation (10,000 IU/day) in D3 insufficient patients (baseline 25-OHD <33ng/ml (82.5 nmol/ml)) patients.

SECONDARY OUTCOMES:
Proportion of participants reaching 25-hydroxycholecalciferol concentration >=33ng/ml (82.5 nmol/ml) between groups | 12 weeks
  To compare the proportion of participants reaching a laboratory "normal" 25-hydroxycholecalciferol concentration >=33ng/ml (82.5 nmol/ml) between D3 supplement groups following 12-weeks of D3 supplementation at 10,000 IU.day
Change in mean Klotho protein concentration | Baseline and 12 weeks
  To explore the expression of Klotho protein, and analytes associated with VitD homeostasis, comparing VitD sufficient, i.e. 25-OHD >=33ng/ml (82.5 nmol/ml), patients to those who are VitD insufficient, i.e. 25-OHD <33ng/ml, at baseline screenings, and to compare Klotho protein expression in VitD insufficient participants before and after D3 supplementation (10,000 IU/day), stratified by supplement group assignment.
Change in Toll-like receptor concentration in monocytes | Baseline and 12 weeks
  To explore the change in IFN-gamma induced TLR-4 expression in human monocytes (ex-vivo), comparing VitD sufficient, i.e. 25-OHD >=33ng/ml (82.5 nmol/ml), patients to those who are VitD insufficient, i.e. 25-OHD <33ng/ml, at baseline screenings, and to compare the change in IFN-gamma induced TLR-4 expression in human monocytes (ex-vivo) between VitD groups, following 12 weeks of supplementation with one of three forms of VitD3: lipid-emulsified, non-emulsified chewable tablet, and a non-emulsified encapsulated form.
Change in mean cardiometabolic risk factors | Baseline- 12 weeks
  To explore change in mean fasting glucose, hemoglobin A1c, total cholesterol, fasting insulin, HOMA-IR, LDL, HDL-C, and triglycerides will be reported following 12-weeks of D3 supplementation (10,000 IU/day) in healthy humans

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Bradley, ND, MPH, Principal Investigator — Bastyr University
Locations (2):
- United States (2):
  - Lokahi Health Center, Kailua-Kona, Hawaii
  - Bastyr University, Kenmore, Washington